CLINICAL TRIAL: NCT00370526
Title: HEmodynamic Assessment of Optimal Left Heart Lead Placement for Heart Failure Enabled by Magnetic Navigation
Brief Title: HEAL-HF: A Cardiac Resynchronization Therapy (CRT) Outcomes Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Stereotaxis (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Mark Jacob, Senrior Manager of Clinical Affairs, Stereotaxis, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM-CLIN 008
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure; resynchronization; CRT; Bi-V pacemaker; LV lead placement; hemodynamic assessment; CRT Outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acute hemodynamic assessment using PV Loops (CD Leycom, The Netherlands) during LV lead placement

SUMMARY:
The literature shows that approximately 40% of individuals who receive a cardiac resynchronization therapy (CRT) device for symptomatic congestive heart failure (CHF) do not have a clinical benefit from the device. The HEAL-HF protocol will compare the outcomes of conventionally placed CRT devices with magnetically placed CRT devices by assessing hemodynamic parameters during the magnetic placement of the left ventricular (LV) lead.

DETAILED DESCRIPTION:
Baseline information will be obtained including QoL, 6-minute walk, and echo measurements. The patient will be randomized to receive a conventionally-placed LV lead or randomized to receive a magnetically-placed LV lead. The magnetic group will have acute hemodynamics assessed during the procedure to evaluate the best response of the left ventricle during pacing. Patients will be followed for 6 months with a re-evaluation of the baseline tests to assess the change in HF symptoms. Adverse events will also be recorded during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiomyopathy
* Ejection Fraction (EF) <= 35%
* QRS duration >= 120 msec
* Standard heart failure (HF) oral medications for at least 1 month
* Evidence of mechanical dyssynchrony
* NYHA Class III or IV

Exclusion Criteria:

* Persistent or chronic atrial fibrillation (AF)
* Hemodynamically unstable or uncontrolled arrhythmias
* Unstable angina
* Aortic valve (AV) insufficiency or stenosis
* Mitral valve (MV) regurgitation > 2+
* Active infection
* Contraindications for heparin
* Dependence on atrial pacing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction in end systolic volume (ESV) | 6 months

SECONDARY OUTCOMES:
New York Heart Association (NYHA) Class | 6 months
6 minute walk | 6 months
Quality of life (QoL) | 6 months
Cardiac-related mortality | 6 months
HF-related hospitalizations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, PhD, Principal Investigator — San Raffaele University Hospital
Locations (5):
- United States (3):
  - Northeast Georgia Heart Center, PC, Gainesville, Georgia
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Virginia - Virginia Commonwealth University, Richmond, Virginia
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada
- San Raffaele University Hospital, Milan, Italy